CLINICAL TRIAL: NCT01492699
Title: Single Site, Open Label Pilot Study of PRX-03140 to Assess Safety for Use in Adult Subjects With Post Traumatic Stress Disorder.
Brief Title: Pilot Study of PRX-03140 to Assess Safety for Use in Adult Subjects With Post Traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-PTSD-NT/001
Record Dates: First submitted 2011-12-09; First posted 2011-12-15 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PRX-03140 (Experimental): PRX-03140 for the treatment of PTSD
  Interventions: Drug: PRX-03140

INTERVENTIONS:
Drug: PRX-03140 — 50 mg PRX-03140 capsules once daily for 2 weeks. After 2 weeks, the dose will increase to 100mg PRX-03140 once daily for 10 weeks.

SUMMARY:
This is a clinical study for adult subjects with Post Traumatic Stress Disorder.

DETAILED DESCRIPTION:
Open label clinical study to evaluate the efficacy of PRX-03140 in reducing PTSD symptoms

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between ages 18-55
2. The subject has signed and dated the written informed consent to participate in the study
3. The subject is able to understand and comply with written and verbal protocol requirements, instructions, and protocol-stated restrictions
4. The subject meets criteria for PTSD as defined by the DSM-IV-TR
5. Stable use of clinically prescribed medications
6. Subject able to complete baseline, 4 weeks, and 12 week psychological and cognitive evaluation
7. Female subjects - not surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) for at least 6 months or at least 2 years postmenopausal - must agree to utilize one of the following forms of contraception, if sexually active with a male partner, from screening through completion of the study. Approved forms of contraception are abstinence, hormonal (oral, implant, transdermal, vaginal, or injection) in use at least 3 consecutive months prior to the first dose of study medication, double barrier (condom with spermicide; diaphragm with spermicide), intrauterine device (IUD), or vasectomized partner (6 months minimum since vasectomy).

Exclusion Criteria:

1. Actively alcohol or drug dependent as defined by DSM-IV-TR Criteria
2. Patient actively suicidal within last 12-months or with current suicidal ideation
3. History of schizophrenia, bipolar disorder, attention deficit hyperactivity disorder, learning disability, stroke, multiple sclerosis or seizure disorder by interview
4. Participation in a clinical drug research study within the past 30 days
5. Subject currently taking any SSRI or anti-depressant medication.
6. Pregnant or breastfeeding females
7. Subjects will be excluded based on lab values, ECG findings, or physical findings that the Investigators deems exclusionary.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in adverse events from baseline | weekly for 4 weeks then every 4 weeks until week 14
  adverse events will be evaluated at every visit

SECONDARY OUTCOMES:
Change from baseline in PTSD and mood related symptoms | weekly for 4 weeks then every 4 weeks until week 14
  subjects will fill out PTSD and mood related symptoms questionnaires at each visit to show any changes in symptoms from baseline

CONTACTS AND LOCATIONS:
Overall Officials: John Abernethy, MD, Study Director — Alachua Government Services, Inc.
Locations (1):
- Sarkis Clinical Trials, Gainesville, Florida, United States